CLINICAL TRIAL: NCT02677831
Title: Healthy Aging Longitudinal Study in Taiwan (HALST)
Brief Title: Healthy Aging Longitudinal Study in Taiwan
Acronym: HALST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other); Hope Doctors Hospital (Unknown); Changhua Christian Hospital (Other); Puzi Hospital (Unknown); Yuan's General Hospital (Other); Mennonite Christian Hospital (Other); CHC Hospital Group (Unknown); Northwestern University (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Chao A. Hsiung, Distinguished Investigator/Director, National Health Research Institutes, Taiwan
Other Study IDs: EC0970608
Record Dates: First submitted 2016-01-24; First posted 2016-02-09 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Diseases; Metabolic Diseases
Keywords: Physical functioning; Neuropsychiatric Disorders; Frailty
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Diseases; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, urine.
Oversight: Data Monitoring Committee: No

SUMMARY:
The general aim of this study is to establish a longitudinal cohort of older persons in order to examine the physiological, environmental and genetic risk factors for physical disability, frailty, cardiovascular disease, and neuropsychiatric disorders in older persons and to examine the benefit of healthy lifestyles. The findings from this study will provide information necessary for the development of effective health policy for aging people.

DETAILED DESCRIPTION:
In the proposed research, investigators plan to conduct a longitudinal study on a cohort of 5,000+ men and women ages 55 years or older to address issues related to healthy aging. The study population consists community-based middle to old aged men and women in the catchment area of 7 hospitals (2 in the north, 2 in the middle, 2 in the south and 1 in the east, about half urban half rural). In this proposed study, investigators will recruit the subjects in the catchment area of the above 7 hospitals and expand data collection to include more interviewer-administered data, physical examinations and blood and urine specimens.

In addition, the cohort will be followed annually for mortality and morbidity and will be re-examined every five years.

For this newly proposed study, in order to systematically address issues related to healthy aging, specific aims are grouped into five inter-related areas of emphasis (five component projects). The five component projects are:

A. Factors that may influence physical functioning and its changes in older persons.

B. The benefit of healthy lifestyles on cardiovascular disease risk profile, quality of life and physical functioning in older persons.

C. Individual and macro-level risk factors of cardiovascular disease in older persons.

D. Neuropsychiatric disorders in the elderly: risk factors and impact on health.

E. Genetic and environmental factors for frailty/successful aging and related chronic diseases in the elderly.

The proposed starting date is on March, 2008. The first nine months will be devoted to the development of protocol, manual of operation, pilot testing, central training, and dress rehearsal. The baseline examination will begin in November, 2008 and will last for 4 years. The examination will consist of three parts, a home visit, a clinic examination and the Heart Rate Variability. The home visit will include interviewer-administered questionnaires (informed consent, contact/follow-up information, sociodemographic data, health condition/medical history, family disease history, physical functioning, geriatric conditions, mental health, cognitive function, social and health environments, lifestyles and quality of life, etc.) and physical assessment (peak flow test, grip strength, and physical performance measures). It is estimated that the home visit will take up to 2 hours. The clinic examination will include urine collection, blood pressure, phlebotomy, Primary Care Evaluation of Mental Disorders (high risk people only), anthropometric measures (body height, weight, and circumference measures of waist and hip), body composition, visual test, clock drawing test, the Digit-Symbol Substitution Test, EKG, Heart Rate Variability (HRV), Ankle Brachial Index(ABI), Dual Energy X-ray Absorptiometry (DXA), physical examination, three mobility tests (single leg stance, timed up and go, and six-minute walk test), and a brief questionnaire. The clinic examination is estimated to take approximate 2.5 to 3 hours. Quality of the data collection will be continuously monitored. Two rounds of Heart Rate Variability (HRV) measurements will be conducted. During each round, the HRV will be measured twice with a total duration of about 40 minutes. Those who have installed pacemakers will be excluded from investigators HRV examination. The first round of HRV test will be conducted during the clinic examination, and the second round will be performed about one week later. It is estimated that about 60 participants will need to be enrolled in the HRV test, and each participant needs to complete four times of HRV measurement. This repeated measurement of HRV will allow us to test whether the reliability of investigators HRV measurement is acceptable with an intraclass correlation coefficient (ICC) of at least 0.6 (α=0.05, 1-β=0.8). The HRV test will be stopped when at least 60 participants are enrolled at Taipei site. The responsible investigators and the co-investigators are experienced in the corresponding areas of research. They have been collaborating successfully on various projects for many years. During the study, the investigators will meet via conference call or face-to-face meeting twice a month to discuss issues related to the examination, quality of data, scientific direction, data analyses and manuscript preparation. The proposed study will provide a unique opportunity to enhance investigators understanding of the cardiovascular disease risk factor profile, physical and mental performance and functioning, frailty, quality of life, and morbidity and mortality in a representative cohort of older people in Taiwan. It will provide an opportunity to assess the effects of healthy lifestyles on the prevention of chronic illnesses, disability, and quality of life in older ages. This study of the effects of healthy lifestyles in middle and older ages on overall health among older persons, as investigators propose, has particular societal relevance given the marked growth in numbers of older persons in the Taiwanese population, and their extensive chronic disease-related morbidity, disability, loss of independence, large health care costs, and mortality. Positive results from this study will inform policy regarding the allocation of resources for promoting healthy lifestyles so that the aging population can compress the onset of morbidity and disability, maintaining high quality of life and reducing health care costs.

ELIGIBILITY:
Inclusion Criteria:

* ages 55 years or older

Exclusion Criteria:

* high transmitted disease (such as scabies, open pulmonary tuberculosis)
* severe illness (such as cancer under treatment)
* diagnosed dementia
* severe illness and being bed-ridden, unable to move
* severe mental disorder, cannot be communicated with（MMSE<16）
* dumbness or hearing impairment, unable to complete the interview
* unsighted completely, unable to complete the interview and test
* < 55 years of age
* Other conditions, such as living in a long-term care facility or being hospitalized

Ages: 55 Years to 104 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investigators plan to conduct a longitudinal study on a cohort of 5,000+ men and women ages 55 years or older to address issues related to healthy aging. The study population consists community-based middle to old aged men and women in the catchment area of 7 hospitals (2 in the north, 2 in the middle, 2 in the south and 1 in the east, about half urban half rural). In this proposed study, investigators will recruit the subjects in the catchment area of the above 7 hospitals and expand data collection to include more interviewer-administered data, physical examinations and blood and urine specimens.
Sampling Method: Probability Sample
Enrollment: 5664 (Actual)
Dates: Start 2008-07; Primary Completion 2013-03 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Independence in daily life assessed by Barthel Index | 20 years
  The Barthel Index will be adapted to assess the ability to cope with 10 items of daily activities. These tasks include feeding, moving from wheelchair to bed, personal toilet, getting on and off the toilet, bathing, walking on a level surface, ascending and descending stairs, dressing, controlling bowel, and controlling bladder. The total score ranges from 0 to 100, with 100 representing full independence in doing daily activities.
Independence in daily life assessed by Lawton-Brody Instrumental Activities of Daily Living (IADL) scale | 20 years
  IADL scale is used to measure a participant's ability to adapt to the environment and consists of 8 tasks: shopping, housekeeping, money management, food preparation, laundry, transportation, use of the telephone, and medications. The total score is from 0 (worst) to 8 (best).
Declined rate of physical performance assessed by peak flow test | 20 years
  The peak flow test, is a measure of lung function, the participant is asked to take a deep breath and blow as fast and hard as possible into the meter at a standing or sitting position. The maximum value in liter per minute of three to five trials of forced expiration is chosen as the peak flow.
Declined rate of physical performance assessed by grip strength | 20 years
  The participant is instructed to use the dominant hand to grip the dynamometer as hard as possible three times. The maximum value in kilograms of three trials is recorded as maximal grip strength.
Declined rate of physical performance assessed by Summary Physical Performance Battery (SPPB) | 20 years
  The SPPB, is a measure of lower extremity function and represents the participant's performance on three performance-based tests: 4-meter timed walk, five chair stands, and balance in three different standing positions side by side, semi-tandem, and full tandem. Participants will receive a score of 0 to 4 for each test. The summary performance score is the sum of scores calculated across the three tests, with 0 representing the worst and 12 the best.
Cardiovascular disease incidence by linking the National Health Insurance Research Database in Taiwan | 20 years
Dementia incidence by linking the National Health Insurance Research Database in Taiwan | 20 years
Overall cancer incidence by linking the National Health Insurance Research Database in Taiwan | 20 years
All cause mortality | 20 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu IC, Chang HY, Hsu CC, Chiu YF, Yu SH, Tsai YF, Shen SC, Kuo KN, Chen CY, Liu K, Lee MM, Hsiung CA. Association between dietary fiber intake and physical performance in older adults: a nationwide study in Taiwan. PLoS One. 2013 Nov 11;8(11):e80209. doi: 10.1371/journal.pone.0080209. eCollection 2013. PMID 24244650
- [Result] Wu IC, Lin CC, Hsiung CA, Wang CY, Wu CH, Chan DC, Li TC, Lin WY, Huang KC, Chen CY, Hsu CC; Sarcopenia and Translational Aging Research in Taiwan Team. Epidemiology of sarcopenia among community-dwelling older adults in Taiwan: a pooled analysis for a broader adoption of sarcopenia assessments. Geriatr Gerontol Int. 2014 Feb;14 Suppl 1:52-60. doi: 10.1111/ggi.12193. PMID 24450561
- [Derived] Tseng HY, Lockenhoff C, Lee CY, Yu SH, Wu IC, Chang HY, Chiu YF, Hsiung CA. The paradox of aging and health-related quality of life in Asian Chinese: results from the Healthy Aging Longitudinal Study in Taiwan. BMC Geriatr. 2020 Mar 5;20(1):91. doi: 10.1186/s12877-020-1446-y. PMID 32138691
- [Derived] Chuang SC, Chen HL, Tseng WT, Wu IC, Hsu CC, Chang HY, Chen YI, Lee MM, Liu K, Hsiung CA. Circulating 25-hydroxyvitamin D and physical performance in older adults: a nationwide study in Taiwan. Am J Clin Nutr. 2016 Nov;104(5):1334-1344. doi: 10.3945/ajcn.115.122804. Epub 2016 Oct 12. PMID 27733394